CLINICAL TRIAL: NCT06808620
Title: The Effect of Using Peanut Balls During Labor on Perceived Labor Pain, Duration, and Self-Efficacy: A Randomized Controlled Study
Brief Title: The Effect of Using Peanuts Balls at Birth
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Funda Citil Canbay, Association Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/295
Record Dates: First submitted 2024-10-11; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Exercise; Labor; Birth
Keywords: Labor Pain; Labor Duration; Self-Sufficiency; Peanut Ball; Vaginal Birth
MeSH Terms: conditions — Motor Activity; Labor Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Control (No Intervention): The group which has no implementation
- Use of peanut ball (Experimental): The group which peanut ball are implemented
  Interventions: Other: The group where the peanut ball is used

INTERVENTIONS:
Other: The group where the peanut ball is used — Before the application, the appropriate ball size for the physical characteristics and comfort of the pregnant women will be determined. Pregnant women will be given 4 different sizes of peanut balls with a diameter of 40, 55, 65 and 75 cm. In order for the pregnant woman to continue her in-bed balance exercises and position changes, she will be allowed to sit on the peanut ball with her knees and hips at an angle of approximately 90° and her spine upright. A 40-55 cm birthing ball will be used for women between 150-160 cm tall, a 65 cm birthing ball for women between 160-170 cm tall, and a 75 cm birthing ball for women between 170-185 cm tall. Position changes with the peanut ball will be carried out in accordance with a position/exercise guide prepared by researchers in line with literature information. The peanut ball will be applied in 6 different positions. These positions to be applied will consist of side-lying positions, semi-sitting pose, forward bending pose and squatting pos
  Other Names: The group which has no implementation
  Arms: Use of peanut ball

SUMMARY:
The necessity of applying the research on humans, whether the application has been done in our country or in other countries before, if it has been done, additional data expected from this study or differences from this study from others, and the expected benefits, please explain within the framework of scientific data.

With this planned study, it is aimed to increase the activities of pregnant women during birth by using peanut balls during the birth process, to support the pregnant women psychologically, to reduce labor pains, to shorten the duration of normal birth, to increase self-efficacy for normal birth, to reduce cesarean section rates, to increase labor satisfaction, to reduce fear of birth, to expand the pelvic diameter, to stretch the pelvic muscles and to provide positive gains on connective tissues. With this planned study, it is aimed to reduce labor pain, to shorten the duration of labor and to increase the self-efficacy of the pregnant women for vaginal birth by using peanut balls during the birth process and benefiting from the stated benefits.

When the literature review was done, it was determined that partial studies were conducted on the effect of peanut balls on birth in Turkey and in the world, and it was determined that peanut balls are not used in delivery rooms in Turkey despite having many benefits on birth. This study aims to pioneer the widespread use of peanut balls in Turkey. This study was planned to determine the effect of using peanut balls on labor duration, perceived labor pain and self-efficacy in primiparous pregnant women with a cervical dilation of 4 cm and above, in line with the vaginal birth plan. The aim of the planned study is to evaluate the effect of changing position with peanut balls during labor on perceived labor pain, labor duration and self-efficacy levels for normal birth.

The hypotheses of the study proposed for this purpose are; H1: Labor pain, duration and self-efficacy of pregnant women who use peanut balls during labor are different from the control group.

H2: Perceived labor pain decreases in pregnant women who use peanut balls during labor compared to the control group.

H3: The duration of labor (the time period from the active phase to the completion of the transition phase) is shortened in pregnant women who use peanut balls during labor compared to the control group.

H4: The duration of labor (the second stage of labor) is shortened in pregnant women who use peanut balls during labor compared to the control group.

H5: Using peanut balls during birth increases the self-efficacy level in pregnant women compared to the control group.

The peanut ball will be applied in 6 different positions. These positions will consist of side-lying positions, half-sitting pose, forward bending pose and squatting positions. The positions to be applied are planned as in-bed. Pregnant women will be informed about the positions to be applied. The peanut ball will be applied for 20-25 minutes and a 5-10 minute break will be given. The introductory and obstetric information form will be filled out once for each patient. The partograph will be started with the start of the peanut ball use and will end with the end of labor. The visual comparison scale (VAS) and the self-efficacy scale for normal labor will be used 3 times in this study. It will be applied when the dilation is 4 cm and below before the application, immediately after the peanut ball application and half an hour after the peanut ball application.

DETAILED DESCRIPTION:
Even if there is no risk, the success of the labor is shaped by the mobility, general well-being and needs of the pregnant woman. While social support is provided in line with the principles of individualized care during labor, positioning the woman in the most comfortable positions positively affects the sense of control during labor. This reduces unnecessary interventions and the possibility of cesarean section during labor. Peanut-shaped birth balls are popular in countries with high vaginal birth rates and among researchers. Reducing labor pain and keeping labor durations at an optimum level is possible with non-pharmacological methods. It has been proven that using peanut balls during labor reduces cesarean section rates, increases maternal satisfaction with perceived labor success, and shortens labor pain and labor duration. Using peanut balls during labor makes it easier for pregnant women to move into different positions safely and comfortably. Despite the known benefits of peanut balls, they are not common in births in Turkey. To our knowledge, although some birth balls are observed to be used during labor, no study has been found testing the perception of self-sufficiency during labor shaped by the perceived labor pain, labor duration and feelings of control of peanut balls during labor. The planned research is a pretest-posttest randomized control group experimental study to examine the effect of using peanut balls during labor on perceived labor pain, duration and self-efficacy. The universe of the research will consist of pregnant women who apply to Hakkari Yüksekova Maternity and Childbirth Hospital for vaginal delivery. The sample of the research was calculated with power analysis. "Descriptive and Obstetric Information Form", "Visual Comparison Scale (VAS)", "Partograph" and "Self-efficacy Scale for Normal Delivery" will be used to collect the data. Different position changes will be applied to the study group with peanut balls during labor. The control group will benefit from the hospital's routine care. The partograph will end with the end of labor. VAS and self-efficacy scale for normal delivery will be used 3 times. Descriptive statistics in the analysis will be applied according to the results obtained from normal distribution tests, parametric or nonparametric tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women should be in their 38-42nd weeks of pregnancy
* Cervical dilation should be 3 cm or more
* Single live baby
* Vertex position should be
* No health problems
* No communication problems
* No risky pregnancies
* Those who can have vaginal birth
* Primiparous pregnancy
* Active phase

Exclusion Criteria:

1. Indication for Caesarean section
2. Complications during delivery
3. Unwilling to continue working
4. Risky pregnancies
5. Pregnant women without inclusion criteria

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Perceived labor pain (Visual Analog Scale) | During labor
  The visual analog scale (VAS) was developed by Price et al. (1983) to determine the level of perceived pain during labor. VAS is used easily and conveniently by converting some situations that are difficult to measure quantitatively into numerical values (Yeşilyurt and Faydalı, 2020). The visual comparison scale is in the form of a 10 cm vertical and horizontal ruler. In order to determine the intensity of pain, one end indicates the lowest level of perceived pain and the other end indicates that the intensity of pain increases. If there is no perceived pain, "0" is shown, and the number "10" indicates the highest level of pain. The pregnant woman in pain evaluates her own pain out of 10 and indicates the appropriate number for herself. A score of 1-4 on this scale indicates mild pain, 5-6 indicates moderate pain, and a score above 7 indicates severe pain (Ayan et al., 2013). No cut-off point is specified in the visual comparison scale. Its use is recommended in comparative studies
Labor duration | Labor
  Effect of using peanut ball on labor duration
Perception of Self-Efficacy for Normal Birth | During labor
  Effect of using peanut ball on self-efficacy perception for normal birth

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Universty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to provide information about plans to share individual participant data (IPD).